CLINICAL TRIAL: NCT05576233
Title: Comparison of Blood Culture Contamination Rates Between the Use of Povidine Iodine/Alcohol for Skin Antisepsis and the Use of Chlorhexidine/Alcohol (ChloraPrep) for Skin Antisepsis: An Open-label, Randomized Controlled Trial
Brief Title: • Comparison of Blood Culture Contamination Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ilker devrim, Professor. Dr., Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: skin antisepsis study
Record Dates: First submitted 2022-10-09; First posted 2022-10-12 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Blood Culture Contamination
Keywords: Blood culture contamination; Chloraprep ( alcohol/ chlorhexidine); Povidine/iodine; Topical disinfectants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.The culture taken after disinfection with providing/iodine (Active Comparator): 1.Blood cultures routinely performed with alcohol/povidine-iodine
  Interventions: Procedure: disinfection of the surface that the blood culture is taken
- 2.The culture taken after disinfection with chlorhexidine/alcohol (Active Comparator): 2. Blood cultures routinely performed with chlorhexidine/alcohol
  Interventions: Procedure: disinfection of the surface that the blood culture is taken

INTERVENTIONS:
Procedure: disinfection of the surface that the blood culture is taken — lood cultures can be routinely performed with alcohol/povidine-iodine or alcohol/chlorhexidine. The topical disinfectants used in the two applications are the topical disinfectants included in the guidelines and currently applied in our hospital.

SUMMARY:
In this study, blood culture contamination rates will be compared in patients who used povidine/iodine-alcohol and chlorhexidine/alcohol, which were applied before the blood culture was taken by randomized two methods routinely used in this study.

DETAILED DESCRIPTION:
Detection of the pathogen in blood cultures as soon as possible reduces mortality significantly by providing timely initiation of treatment1. However, when skin antisepsis is not performed properly, an increase in the rate of contamination is observed. In this study, it was planned to compare the contamination rate of two antiseptics, povidine iodine/alcohol and Chlorhexidine/alcohol used as skin antisepsis, in the blood culture taken.

Full randomization" will be applied in the study. Multiples of 3 of the patients to be included in the study will be included in the "Chloraprep" group, the remaining patients and multiples of 2 will be included in the "povidine/iodine" group. . According to the number of samples determined for each institution, patients who came to the outpatient clinic during data collection and accepted to participate in the study will be randomly selected.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be hospitalized at SBU Izmir Dr. Patients who are hospitalized in the Pediatric Infection Service of Behçet Uz Pediatrics and Surgery Training and Research Hospital, and who will require blood culture indications will participate in the study If they are willing to

Exclusion Criteria:

* The patents with central lines will be excluded.
* The patient who were transferred from ICU's will be excluded.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood Contamination | 14 days
  The primary endpoint of the study was to reduce the rate of contamination in blood cultures.